CLINICAL TRIAL: NCT00593463
Title: Drug Discrimination in Methadone-Maintained Humans Study 1
Acronym: OMDD1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Alison Oliveto, Ph.D./Principal Investigator, University of Arkansas for Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Double
Other Study IDs: R01DA010017-01 (NIH); 57184; R01DA010017 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Drug Dependence
Keywords: opioid dependence; methadone; opioid
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders | interventions — Cycloserine; Verapamil; Diltiazem; Gabapentin; Isradipine; Naloxone; Nifedipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Receives 2-4 of the interventions listed
  Interventions: Drug: Cycloserine; Drug: Diltiazem; Drug: Gabapentin; Drug: Isradipine; Drug: Naloxone; Drug: Nifedipine; Drug: Placebo; Device: Saline; Drug: Verapamil

INTERVENTIONS:
Drug: Cycloserine — Cycloserine: 500, 675, 750 mg oral capsule may possibly be given
  Other Names: Calan; Veralan
Drug: Diltiazem — Diltiazem: 30, 60, 120 mg oral capsule may possibly be
  Other Names: Cardizem
Drug: Gabapentin — Gabapentin: 100, 200, 400 mg oral capsule may possibly be given
  Other Names: Neurontin
Drug: Isradipine — Isradipine: 5, 10 mg oral capsule may possibly be given
  Other Names: DynaCirc
Drug: Naloxone — Naloxone: 0.15 mg/70 kg or 0.2 mg I.M. injection may possibly be given
  Other Names: Narca
Drug: Nifedipine — Nifedipine: 5, 10, 20 mg oral capsule may possibly be given
  Other Names: Adalat; Procardia
Drug: Placebo — Placebo (sugar pill or microcrystalline cellulose): oral capsule may possibly be given
Device: Saline — Saline: I.M. injection may possibly be given
Drug: Verapamil — Verapamil: 30, 60, 120 mg oral capsule may possibly be given
  Other Names: Veralan

SUMMARY:
This study involves giving psychoactive drugs intramuscularly (injected into the muscle of the upper arm or the hip) and/or orally, and measuring the subject's ability to tell the difference between one drug and another, as well as measuring the effects of the drugs on mood, physiology (e.g., heart rate, blood pressure, respiration rate) and behavior. Each subject will receive 2-4 of the listed interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 18-65.
2. Participation in the UAMS Substance Abuse Treatment Clinic Methadone Maintenance Program or the CATAR Clinic Little Rock with maintenance on a stable dose of methadone (+ or - 10 mg) for at least 1 month prior to study entry.
3. Subjects would have to be in "good standing" in the methadone maintenance program in order to participate; i.e., compliance with scheduled medication and group therapy session hours. This would be defined as < 3 missed methadone medications and missed < 3 group or <3 individual therapy sessions in the two months prior to study participation
4. Subjects must submit a urine sample negative for illicit drugs prior to study entry.
5. Subjects must be able to read and understand English.

Exclusion Criteria:

Exclusion criteria

1. Ill health (major cardiovascular, renal, endocrine, hepatic disorder, to be determined by history provided by the prospective subject or laboratory evaluation as outlined below).
2. Current diagnosis of other drug or alcohol physical dependence (other than tobacco).
3. History of major psychiatric disorder (psychosis, schizophrenia, bipolar, depression)
4. Pregnancy, plans to become pregnant or inadequate birth control.
5. Present or recent use of over-the-counter psychoactive drug, prescription psychoactive drug or drug that would have major interaction with drugs to be tested.
6. History of severe reaction to Narcan challenge, which may have been given as part of admission into the Methadone Maintenance Program or to reverse overdose.
7. Liver function tests greater than 3 times normal, BUN and Creatinine outside normal range, or thyroid function tests outside normal range.
8. EKG abnormalities including but not limited to: bradycardia (<60 bpm); prolonged with QTc interval (>420 msec); Wolff-Parkinson White syndrome; wide complex tachycardia; 2nd degree, Mobitz type II heart block; 3rd degree heart block; left or right bundle branch block.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Drug Discrimination Measure | Every session

SECONDARY OUTCOMES:
Self-reported effects | Every Session
Vital Signs | Every session

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States